CLINICAL TRIAL: NCT05360186
Title: The Efficacy and Safety of a New Cross-linked Hyaluronan Gel to Prevent Adhesion After Ultrasound-guided Manual Vacuum Aspiration (USG-MVA): A Prospective Randomized Controlled Trial
Brief Title: New Cross-linked Hyaluronan Gel to Prevent Adhesion After USG-MVA: RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Health and Medical Research Fund (Other Government)
Responsible Party: Principal Investigator, Chung Pui Wah Jacqueline, Associate Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2021.702-T
Record Dates: First submitted 2022-03-31; First posted 2022-05-04 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: First Trimester Abortion; Surgical Abortion; Miscarriage With Afibrinogenemia
Keywords: First Trimester Abortion; Surgical Abortion; Intrauterine adhesion; Hyaluronan gel; Protective Agents; Hyaluronic Acid; Manual vacuum aspiration; Miscarriage
MeSH Terms: conditions — Gynatresia; Abortion, Spontaneous

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Group A): NCH gel after USG-MVA (Experimental): In the intervention group (Group A), a 15 cm sterile delivery cannula will be inserted through the internal os and a syringe of NCH gel (5ml) will be applied to the uterine cavity after cleansing the cervix with an antiseptic solution.
  Interventions: Device: MateRegen® gel (BioRegen)
- Controlled group (Group B): No NCH gel after USG-MVA (No Intervention): In the control group (Group B), as the patient is conscious during the procedure, an empty 5ml syringe will be inserted into the internal os and held for 1 minute as a sham procedure.

INTERVENTIONS:
Device: MateRegen® gel (BioRegen) — Modification of Hyaluronic acid structure to 3-dimensional self-cross-linked network structure enables all-dimensional coverage of tissue surface to enhance better healing process. Self-cross-linked HA hydrogels can maintain the biocompatibility and biodegradability that characterize the unmodified material. Moreover, high dynamic viscosity enables continuous indwelling in the uterine cavity. The gel could provide precise regulation, and degradation and absorption time prolonged to 7-14 days post operatively, which completely cover key postoperative healing period (5-7 days), at the highest time of intrauterine adhesion formation.
  Arms: Intervention group (Group A): NCH gel after USG-MVA

SUMMARY:
The objective of this prospective, randomized controlled study was to evaluate the effectiveness of this NCH gel in the prevention of IUA development as assessed by hysteroscopy after USG-MVA, in the treatment for first-trimester miscarriage.

* To study the severity and extent of the IUA as assessed by the AFS and ESGE adhesion score in both groups of patients.
* To examine the rate of complications or side effects with the NCH gel.
* To assess the subsequent menstrual history and reproductive outcome in both groups of patients.

DETAILED DESCRIPTION:
There is limited data to evaluate the incidence of IUA after using this NCH gel in patients undergoing surgical evacuation via USG-MVA for the treatment of first-trimester miscarriage. Previous RCT showed a significant reduction in IUA with the use of NCH gel, with IUA detected in only 9.5% of patients with NCH gel applied compared to 24.1% in the control group. However, the group did not involve patients undergoing surgical evacuation by USG-MVA.

Therefore, the objective of this prospective, randomized controlled study was to evaluate the effectiveness of this NCH gel in the prevention of IUA development as assessed by hysteroscopy after USG-MVA, in the treatment of first-trimester miscarriage.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years old or above
* No previous history of IUA/ Asherman's syndrome
* No previous surgical history of EVA or dilatation or curettage or surgical termination of pregnancy or caesarean section
* No previous history of therapeutic hysteroscopic surgeries
* Voluntary informed consent and understanding of study

Exclusion Criteria:

* previous therapeutic hysteroscopic procedures (e.g. endometrial ablation, removal of fibroids or polyps, surgical correction of congenital uterine anomalies or adhesiolysis)
* suspicion of molar pregnancy
* genital tract malformation
* suspicion of active infection or genital tract malignancy or genital tuberculosis
* abnormal blood coagulation
* inability to tolerate pelvic examination known
* suspected intolerance of hypersensitivity to NCH gel or its derivatives
* patient refusal

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-06-14 (Actual); Primary Completion 2026-05-14 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of IUA | 8-12 weeks after MVA
  To determine the incidence of IUA or after USG-MVA for the treatment of first-trimester miscarriage in both intervention and control groups.

SECONDARY OUTCOMES:
Severity and extent of the intrauterine adhesions as assessed by the AFS adhesion score | 8-12 weeks after MVA
  To study the severity and extent of the intrauterine adhesions as assessed by the AFS adhesion score in both groups of patients.
  The American Fertility Society's (AFS) classification of intrauterine adhesions:
  Stage I (mild) with score 1-4, Stage II (moderate) with score 5-8, Stage III (severe) with score 9-12
Severity and extent of the intrauterine adhesions as assessed by the ESGE adhesion score | 8-12 weeks after MVA
  To study the severity and extent of the intrauterine adhesions as assessed by the European Society of Gynaecological Endoscopy (ESGE) adhesion score in both groups of patients. It includes grades I and II as mild adhesion, grade III as moderate adhesion, grades IV and V as severe adhesion
Complications or side effects with the NCH gel. | 8-12 weeks after MVA
  To examine the rate of complications or side effects with the NCH gel.
Subsequent menstrual frequency | 8-12 weeks after MVA
  To assess the subsequent menstrual frequency in both groups of patients. Frequency - average 28 days <24 days Frequent, >38 days Infrequent Frequency - average 28 days <24 days Frequent, >38 days Infrequent
Subsequent reproductive outcome | 8-12 weeks after MVA
  To assess the rate of pregnancy in both groups of patients

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No